CLINICAL TRIAL: NCT02984384
Title: PREVENTion of Clot in Orthopaedic Trauma (PREVENT CLOT): A Randomized Pragmatic Trial Comparing the Complications and Safety of Blood Clot Prevention Medicines Used in Orthopaedic Trauma Patients
Brief Title: PREVENTion of Clot in Orthopaedic Trauma
Acronym: PREVENT CLOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PCS-1511-32745
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Blood Clot; Trauma
Keywords: Trauma; Blood clot; Venous Thromboembolism; Pulmonary Embolism; Deep Vein Thrombosis; Thromboprophylaxis; Blood clot prevention; trauma patients
MeSH Terms: conditions — Thrombosis; Wounds and Injuries; Venous Thromboembolism; Pulmonary Embolism; Venous Thrombosis | interventions — Aspirin; Heparin, Low-Molecular-Weight; Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Molecular Weight Heparin (LMWH)-Enoxaparin (Active Comparator): Injection of 30 mg enoxaparin, twice a day via injection
  Interventions: Drug: Low Molecular Weight Heparin (LMWH)
- Acetylsalicylic acid (ASA)-Aspirin (Active Comparator): Enteral ingestion or administration of 81 mg ASA, twice a day
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Acetylsalicylic acid — The Aspirin intervention will be 81 mg enteral (by mouth, feeding tube or rectal) twice a day with no variation in dosing allowed.
  Other Names: Aspirin
  Arms: Acetylsalicylic acid (ASA)-Aspirin
Drug: Low Molecular Weight Heparin (LMWH) — The LMWH intervention will be 30 mg enoxaparin subcutaneous (under the skin) twice a day with variations in dosing allowed, per the standard of care at sites, as needed for patients who are very obese or exhibit renal dysfunction.
  Other Names: Enoxaparin
  Arms: Low Molecular Weight Heparin (LMWH)-Enoxaparin

SUMMARY:
The purpose of this study is to compare aspirin versus low-molecular weight heparin (LMWH) (Enoxaparin) as a thromboprophylaxis in patients who sustain a fracture.

DETAILED DESCRIPTION:
Patients who sustain orthopaedic trauma are at an increased risk of venous thromboembolism (VTE), including fatal pulmonary embolism (PE). Current guidelines recommend low-molecular-weight heparin (LMWH) for VTE prophylaxis in orthopaedic trauma patients. However, emerging literature in total joint arthroplasty patients suggests the potential clinical benefits of VTE prophylaxis with aspirin. This trial aims to determine if aspirin is non-inferior to LMWH for thromboprophylaxis in fracture patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a planned operative or non-operative pelvis or acetabular fracture, or any operative extremity fracture proximal to the metatarsals or carpals.
* Patients at increased risk of blood clot(s) from their orthopaedic injury(ies) and will receive prophylactic blood thinner regimen per standard of care.
* Patients 18 years or older.

Exclusion Criteria:

* Patients who present to the hospital more than 48 hours post injury
* Patients who received more than 2 doses of LMWH or aspirin for initial VTE prophylaxis
* Patients on long term blood thinners (other than low-dose aspirin or platelet inhibitors such as Plavix or Aggrenox)
* Patients who have had a VTE within the last 6 months
* Patients on therapeutic (as opposed to prophylactic) blood thinners for an acute issue at the time of admission
* Patients who have a newly diagnosed indication for therapeutic blood thinners (for example vascular injury) that will require therapeutic anticoagulation for more than one week
* Patients who cannot receive either of the study medications due to an allergy (history of heparin induced thrombocytopenia, allergy to aspirin, or NSAIDs) or other medical contraindication to blood thinners
* Patients who are on higher dose aspirin (>81 mg once a day or higher) for medical reasons or who will be treated with higher dose aspirin
* Patients with underlying chronic clotting disorders (i.e. Factor V Leiden, hyperhomocysteinemia, Protein C and S deficiency) that require full dose anticoagulation or are a contraindication to venous thromboembolism chemoprophylaxis
* Patients with end stage renal disease or impaired creatinine clearance <30 ml/min at time of randomization(note: creatinine clearance does not need to be documented if prescribing physician would order medication without test as SOC)
* Pregnant or lactating patients
* Prisoners
* Patients who do not speak either English or Spanish
* Patients who are likely to have severe problems maintaining follow-up
* Patients, based upon the clinical judgment of the treating clinician, NOT equally suited for treatment with either aspirin or low-molecular-weight heparin
* Patients may be excluded for other reasons at the discretion of the treating physician; the reason for exclusion must be documented on the screening form
* Patients who have a known COVID-19 diagnosis prior to fracture treatment or within 3 months of the index fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12424 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert O'Toole, MD, Principal Investigator — University of Maryland; Renan Castillo, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Tara Taylor, MPH, Study Director — Johns Hopkins Bloomberg School of Public Health; Katherine Frey, PhD, MPH, RN, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (21):
- United States (19):
  - University of Arizona, Tucson, Arizona
  - University of Miami Ryder Trauma Center, Miami, Florida
  - Methodist Hospital, Indianapolis, Indiana
  - University of Maryland R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Brown University, Providence, Rhode Island
  - University of Tennessee, RegionOne Medical Center, Memphis, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas
  - San Antonio Military Medical Center, San Antonio, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Harborview Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Canada (2):
  - University of Calgary, Foothills Medical Centre, Calgary, Alberta
  - McMaster University, Hamilton General Hospital, Hamilton, Ontario

REFERENCES:
- [Background] O'Toole RV, Stein DM, Frey KP, O'Hara NN, Scharfstein DO, Slobogean GP, Taylor TJ, Haac BE, Carlini AR, Manson TT, Sudini K, Mullins CD, Wegener ST, Firoozabadi R, Haut ER, Bosse MJ, Seymour RB, Holden MB, Gitajn IL, Goldhaber SZ, Eastman AL, Jurkovich GJ, Vallier HA, Gary JL, Kleweno CP, Cuschieri J, Marvel D, Castillo RC; METRC. PREVENTion of CLots in Orthopaedic Trauma (PREVENT CLOT): a randomised pragmatic trial protocol comparing aspirin versus low-molecular-weight heparin for blood clot prevention in orthopaedic trauma patients. BMJ Open. 2021 Mar 24;11(3):e041845. doi: 10.1136/bmjopen-2020-041845. PMID 33762229
- [Derived] Major Extremity Trauma Research Consortium (METRC); O'Toole RV, Stein DM, O'Hara NN, Frey KP, Taylor TJ, Scharfstein DO, Carlini AR, Sudini K, Degani Y, Slobogean GP, Haut ER, Obremskey W, Firoozabadi R, Bosse MJ, Goldhaber SZ, Marvel D, Castillo RC. Aspirin or Low-Molecular-Weight Heparin for Thromboprophylaxis after a Fracture. N Engl J Med. 2023 Jan 19;388(3):203-213. doi: 10.1056/NEJMoa2205973. PMID 36652352
- [Derived] O'Hara NN, Degani Y, Marvel D, Wells D, Mullins CD, Wegener S, Frey K, Joseph T, Hurst J, Castillo R, O'Toole RV; PREVENT CLOT Stakeholder Committee. Which orthopaedic trauma patients are likely to refuse to participate in a clinical trial? A latent class analysis. BMJ Open. 2019 Oct 11;9(10):e032631. doi: 10.1136/bmjopen-2019-032631. PMID 31604788

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Molecular Weight Heparin (LMWH)-Enoxaparin | Acetylsalicylic Acid (ASA)-Aspirin
Started | 6209 | 6215
Completed | 6110 | 6101
Not Completed | 99 | 114

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Molecular Weight Heparin (LMWH)-Enoxaparin | Acetylsalicylic Acid (ASA)-Aspirin | Total
Number analyzed (Participants) | 6110 | 6101 | 12211
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (17.6) | 44.5 (18.0) | 44.6 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2341 | 2269 | 4610
  Male | 3769 | 3832 | 7601
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 736 | 774 | 1510
  Not Hispanic or Latino | 5374 | 5327 | 10701
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 44 | 55 | 99
  Asian | 79 | 82 | 161
  Native Hawaiian or Other Pacific Islander | 14 | 11 | 25
  Black or African American | 1243 | 1264 | 2507
  White | 4197 | 4158 | 8355
  More than one race | 68 | 61 | 129
  Unknown or Not Reported | 465 | 470 | 935
Median body-mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 27.5 [23.8 to 32.8] | 27.1 [23.6 to 31.8] | 27.4 [23.7 to 32.3]
Without Health Insurance [Count of Participants; unit: Participants] | 1288 | 1355 | 2643
Injury Severity Score [Median (Inter-Quartile Range); unit: Scores on a scale] — The injury severity score (ISS) provides an overall score for patients with multiple injuries. Each injury is assigned an abbreviated injury scale (AIS) score and is allocated to one of six body regions. The AIS of the three most severely injured body regions are used produce the ISS score. The ISS is scored between 0 to 75. Scores values as follows: <9 = Mild, 9 - 15 =Moderate, 16-24 = Severe, >/=25 = Profound. Major trauma is considered when ISS> 15.
  Scores on a scale | 9 [4 to 10] | 9 [4 to 10] | 9 [4 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-cause Mortality
Description: Death from any cause
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Molecular Weight Heparin (LMWH)-Enoxaparin | Acetylsalicylic Acid (ASA)-Aspirin
Number analyzed (Participants) | 6110 | 6101
Participants | 45 | 47

2. Secondary Outcome: Number of Participants With Cause-specific Death
Description: Cause specific death. Some participants are reported twice if reason for death met more than one category.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Molecular Weight Heparin (LMWH)-Enoxaparin | Acetylsalicylic Acid (ASA)-Aspirin
Number analyzed (Participants) | 6110 | 6101
Participants
  Death related to PE | 5 | 4
  Death possibly related to PE *includes Death related to PE participants | 14 | 18
  Death unlikely to be related to PE | 31 | 29

3. Secondary Outcome: Non-fatal Pulmonary Embolism
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Molecular Weight Heparin (LMWH)-Enoxaparin | Acetylsalicylic Acid (ASA)-Aspirin
Number analyzed (Participants) | 6110 | 6101
Participants | 90 | 90

4. Secondary Outcome: Deep Vein Thrombosis
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Molecular Weight Heparin (LMWH)-Enoxaparin | Acetylsalicylic Acid (ASA)-Aspirin
Number analyzed (Participants) | 6110 | 6101
Participants | 103 | 151

5. Secondary Outcome: Bleeding Complication
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Molecular Weight Heparin (LMWH)-Enoxaparin | Acetylsalicylic Acid (ASA)-Aspirin
Number analyzed (Participants) | 6110 | 6101
Participants | 869 | 834

6. Secondary Outcome: Wound Complication
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Molecular Weight Heparin (LMWH)-Enoxaparin | Acetylsalicylic Acid (ASA)-Aspirin
Number analyzed (Participants) | 6110 | 6101
Participants | 14 | 8

7. Secondary Outcome: Deep Surgical Site Infection
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Molecular Weight Heparin (LMWH)-Enoxaparin | Acetylsalicylic Acid (ASA)-Aspirin
Number analyzed (Participants) | 6110 | 6101
Participants | 93 | 103

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Low Molecular Weight Heparin (LMWH)-Enoxaparin | Acetylsalicylic Acid (ASA)-Aspirin
All-Cause Mortality (participants affected / at risk) | 45/6110 | 47/6101
Serious Adverse Events (participants affected / at risk) | 260/6110 | 324/6101
Other Adverse Events (participants affected / at risk) | 879/6110 | 840/6101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Molecular Weight Heparin (LMWH)-Enoxaparin (N=6110) | Acetylsalicylic Acid (ASA)-Aspirin (N=6101)
Cardiac arrest (Cardiac disorders) | 3 | 2
General Disorders (General disorders) | 7 | 9 — Other medical disorders
Deep Surgical Site Infections (Infections and infestations) | 93 | 103
Pulmonary Embolism (Blood and lymphatic system disorders) | 90 | 90
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 103 | 151
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Molecular Weight Heparin (LMWH)-Enoxaparin (N=6110) | Acetylsalicylic Acid (ASA)-Aspirin (N=6101)
Wound complication (Injury, poisoning and procedural complications) | 14 | 8
Bleeding complication (Injury, poisoning and procedural complications) | 869 | 834

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT02984384/Prot_SAP_ICF_000.pdf